CLINICAL TRIAL: NCT06895564
Title: A Pilot Study of Proton Stereotactic Body Radiotherapy for Spinal Metastasis
Brief Title: Proton SBRT for Spinal Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Sibley Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2463; IRB00441921 (Other: JHM IRB)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Spinal Metastasis
Keywords: Proton SBRT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Proton SBRT (Other): Proton SBRT for nonhematologic spinal metastasis in patients with complex lesions that are unable to be effectively treated with standard of care photon SBRT.
  Interventions: Radiation: Spinal Proton SBRT

INTERVENTIONS:
Radiation: Spinal Proton SBRT — Patients will be treated with spinal proton SBRT over 5 fractions, with a prescription dose of 6 Gray equivalent (GyE) per fraction to the planning target volume.

SUMMARY:
This is a single-arm pilot study of proton stereotactic body radiotherapy (SBRT) for nonhematologic spinal metastasis in patients with complex lesions that are unable to be effectively treated with standard of care photon SBRT defined as inability to develop a photon SBRT plan that achieves adequate coverage (≥80% planning treatment volume (PTV) coverage)) with a prescription dose of 30 Gy in 5 fractions.

DETAILED DESCRIPTION:
Spine metastases are common with a prevalence of up to 30-50% among patients with a cancer diagnosis. As cancer survivorship improves, durable local control is essential to decrease the risk of pain and neurologic deficits that are associated with spinal metastasis. SBRT for these tumors has demonstrated overall local control rates of approximately 80-90% in the largest published series.

Emerging data highlight the importance of dose escalation for local control in SBRT for spinal metastases. The spinal cord is often the dose limiting structure in patients with spinal metastasis; however, achieving sufficiently high dose and acceptable target coverage while meeting dose constraints of other organs at risk (OARs) such as the small bowel or kidneys also poses a significant technical challenge when using current SBRT modalities for complex cases (e.g., extensive paraspinal disease, epidural disease, disease abutting the kidneys, re-irradiation setting). Maintaining safety is the first priority such that complex cases in current practice often require significant target volume under-coverage in order to meet organ at risk dose constraints, increasing the risk of progression and its associated neurologic morbidity and mortality.

To attempt to improve OAR sparing, proton SBRT has been utilized in other disease sites including prostate, non-small cell lung cancer, and liver. The unique qualities of proton beam therapy may improve target coverage while maintaining OAR sparing in cases where current practice with photon SBRT would require a limited dose and/or under-coverage of the target, both of which are associated with an increased risk of tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof or unequivocal cytologic proof of nonhematologic malignancy. This may be obtained from either the primary or any metastatic site.
2. Participants must have radiographic evidence of spinal metastasis on MRI.
3. Participants must have a complex case that is unable to be effectively treated with photon SBRT, defined as inability to develop a photon SBRT plan that achieves adequate coverage (≥80% PTV coverage) with a prescription dose of 30 Gy in 5 fractions. Such cases include:

   1. Extensive paraspinal disease
   2. Reirradiation setting
   3. Epidural extension (Bilsky grade ≥1c)
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky >60%).
6. Patients of childbearing potential (male or female) must practice adequate contraception due to possible harmful effects of radiation therapy on an unborn child.
7. Patients must have the ability to understand and the willingness to sign a written informed consent document.
8. All patients must be informed of the investigational nature of this study and must be given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Participants may not have a spinal metastases case amenable to standard of care photon SBRT planning techniques that achieve ≥80% PTV coverage with a prescription dose of 30 Gy in 5 fractions.
2. Patients who are unable to receive MRIs will be excluded from the study since MRIs will be critical in treatment planning.
3. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Rate of successful delivery of at least one fraction for 8 of 12 patients with spine metastases | Completion of SBRT treatment, approximately 3 weeks
  To assess the feasibility of proton SBRT in patients with nonhematologic spine metastases that are unable to be effectively treated with photon SBRT. Feasibility will be determined by a successful delivery of at least one fraction for 8 of 12 patients with spine metastases.

SECONDARY OUTCOMES:
Rate of neurologic toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Within 12 months post completion of SBRT treatment
  To estimate the rate of neurologic toxicity, defined as CTCAE v5.0 ≥ grade 3, within 12 months after completion of SBRT.
Interfraction and intrafraction setup and positioning as assessed by motion monitoring | Completion of SBRT treatment, approximately 3 weeks
  To verify inter- and intrafraction patient setup and motion uncertainty as assessed by motion monitoring within 2 millimeters (mm) of patient setup used for radiation planning
Actual spinal cord dose meets dose constraints as recommended by AAPM TG101 | Completion of SBRT treatment, approximately 3 weeks
  To determine whether the actual relative biologic effectiveness (RBE) weighted dose delivered to the spinal cord during proton spinal SBRT meets dose constraints as recommended by American Association of Physicists in Medicine Task Group 101 (AAPM TG101).
Local control rate post-SBRT | 3, 6, 9, and 12 months post-SBRT treatment
  To estimate the local control rate at 3, 6, 9, and 12 months following proton spinal SBRT. Assessed using standard of care imaging obtained every 3 months- comparing imaging studies before SBRT with progressive disease on CT and/or MRI in the treatment volume or at the margin of the treatment field.
Incidence of vertebral compression fracture (VCF) post-SBRT | 3, 6, 9, and 12 months post-SBRT treatment
  To estimate the incidence of VCF within or one vertebra adjacent to the radiation field at 3, 6, 9, and 12 months following proton spinal SBRT. Assessed using standard of care imaging obtained every 3 months up to 12 months- comparing new vertebral body height loss or progression of existing fracture prior to local progression on CT and/or MRI.
Brief Pain Index (BPI) patient-reported outcome pre-SBRT and post-SBRT | Prior to SBRT treatment, and at 3, 6, 9, and 12 months post-SBRT treatment
  To describe patient-reported pain assessments before SBRT and at follow-up evaluations after proton spinal SBRT. Patient-reported pain will be measured using BPI. The score range for BPI is 0-10; a lower score suggests less pain and/or less interference with daily activities.
EORTC Quality of Life (QLQ) BM22 patient-reported outcome pre-SBRT and post-SBRT | Prior to SBRT treatment, and at 3, 6, 9, and 12 months post-SBRT treatment
  To describe patient-reported quality of life (QoL) assessments before SBRT and at follow-up evaluations after proton spinal SBRT. Patient-reported quality of life using the European Organization for Research and Treatment of Cancer bone metastases module (EORTC QLQ-BM22). The score range for EORTC QLQ-BM22 is 0-100; a lower score generally indicates a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States